CLINICAL TRIAL: NCT02866721
Title: A Phase I, Single Center, Open Label, Single Dose, Dose Escalation Study Assessing the Safety and Tolerability of AllogeneiC MEsenchymAl Stem CEll Infusion in Adults With Cystic Fibrosis-CEASE CF
Brief Title: Safety and Tolerability Study of Allogeneic Mesenchymal Stem Cell Infusion in Adults With Cystic Fibrosis
Acronym: CEASE-CF
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Case Western Reserve University (Other); Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Protocol CF-MSC-01; DASENB15A0 (Other Grant/Funding Number: Cystic Fibrosis Foundation Therapeutics)
Record Dates: First submitted 2016-08-07; First posted 2016-08-15 (Estimated); Results first posted 2023-01-30 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Cystic Fibrosis
Keywords: Human Mesenchymal Stem Cells
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Human Allogeneic Mesenchymal Stem Cells (Experimental): One time intravenous (IV) Infusion of up to 5 x 10^6 allogeneic human mesenchymal stem cells per kilogram of body weight (hMSCs/kg). A dose escalation using the "3+3" design will be employed. The three doses are 1 x 10^6, 3 x 10^6, and 5 x 10^6 hMSCs/kg. There is no placebo group. All study participants will receive stem cells.
  Interventions: Biological: Mesenchymal Stem Cells

INTERVENTIONS:
Biological: Mesenchymal Stem Cells — A single dose, one time infusion (in the vein) of one of the following doses of human mesenchymal stem cells (hMSCs): 1 x 10^6, 3 x 10^6 or 5 x 10^6 human mesenchymal stem cells per kilogram body weight (hMSCs/kg) during Visit 2. A traditional 3+3 design will be utilized.
  Allogeneic mesenchymal stem cells (MSCs) will be derived from bone marrow aspirates from a healthy donor whose serum tests negative for cytomegalovirus (CMV) antibodies. Healthy donors will undergo tests for infectious disease and screening for 41 common cystic fibrosis transmembrane conductance regulator (CFTR) mutations. In addition, the MSCs will be validated for in vitro and in vivo efficacy and potency using the in vivo murine pre-clinical model of cystic fibrosis lung infection and inflammation.
  Other Names: MSCs

SUMMARY:
This study is being done to test if it is safe to give stem cells to adult patients with Cystic Fibrosis (CF). The kind of stem cells we are studying are called allogeneic human mesenchymal stem cells or MSCs. MSCs are cells in the body that can grow into different types of cells and respond to various environmental situations. Allogeneic means the cells come from another person (a donor).

This study is only looking at whether or not it is safe to give the stem cells to adults with CF and how the infusion is tolerated. In the future, other studies may be done to see if stem cells can be a new therapeutic treatment for CF.

Stem cells, like other medical products that are intended to treat, cure or prevent disease, generally require approval from the U.S. Food and Drug Administration (FDA) before they can be marketed. The FDA has not approved any stem cell-based products for usual medical care, other than some specific blood forming stem cells for certain indications.

DETAILED DESCRIPTION:
This will be a prospective, single-center, dose-escalation, open-label interventional study to evaluate the safety and tolerability of allogeneic human mesenchymal stem cells (hMSCs) in 15 clinically stable subjects with cystic fibrosis (CF) age ≥ 18 years. After a two to six week screening period, subjects will have a Baseline visit (Days 1-2) where they will undergo a single intravenous infusion of up to 5 x 10E6 allogeneic hMSCs/kilogram (hMSCs/kg) of body weight. Infusions will be performed in the Dahms Clinical Research Unit (DCRU) of University Hospitals Cleveland Medical Center. Subjects will be monitored for any infusion related toxicities for 24 hours after the infusion. Subsequent study visits will occur on Days 7, 14, 28, Months 3 and 6 and telephone calls will occur on Days 4 (or 5), 21, 56 and Month 12. Subject safety and tolerability of a single dose of hMSCs will be evaluated at study visits by review of subject diaries, interval history, pulmonary exacerbations, physical examination, spirometry, and analysis of safety laboratories. Special attention will be placed upon detecting pulmonary exacerbations because anti-inflammatory therapies theoretically could suppress the immune system to the point where it leads to increased infectious complications, although MSC therapeutics are proposed to be antimicrobial. In addition to evaluating safety, this study will also explore efficacy end-points for future clinical trials of MSCs in CF including inflammatory biomarkers from blood and sputum. Serum markers (calprotectin, myeloperoxidase (MPO), granulocyte-macrophage colony-stimulating factor (GM-CSF), interleukin-1β (IL-1β), IL-6, IL8, IL-17, and tumor necrosis factor-a (TNF-a) and sputum markers (white cell counts and differentials, IL-1β, IL-6, IL-8, IL-10, IL-17, GM-CSF, macrophage inflammatory protein-3a (MIP- 3a), TNF-a, and active proteases including neutrophil elastase, alpha-1-antitrypsin, and matrix metallopeptidase 9 (MMP-9) will be determined at Baseline and on Days 7 and 28 for with-in subject comparison. All subject samples will be archived for future projects. Finally, a diagnostic bone marrow exam will be performed on subjects with CF who consent to undergo this optional procedure. Bone marrow samples will be banked and used for future translational studies.

ELIGIBILITY:
Cystic Fibrosis (CF) Subject Inclusion Criteria:

1. Male or female ≥18 years of age
2. Confirmed diagnosis of CF as evidenced by 1 or more clinical features consistent with the CF phenotype and 1 or more of the following criteria:

   1. Sweat chloride equal to or greater than 60 milliequivalents per liter (mEq/L) by quantitative pilocarpine iontophoresis test (QPIT)
   2. 2 well-characterized, disease causing mutations in the cystic fibrosis transmembrane conductance regulator (CFTR) gene
3. Clinically stable with no significant changes in health status within 2 weeks prior to screening.
4. Forced expiratory volume in the first second (FEV1) ≥ 40% predicted for age based on the global lung function initiative equations at the screening visit
5. Weight ≥ 40 kilograms at the screening visit
6. Able to perform repeatable, consistent efforts in pulmonary function testing
7. Written informed consent obtained from the subject.

CF Subject Exclusion Criteria:

1. Use of an investigational agent within the 4-week period prior to Visit 1 (Day -42 to -10)
2. Chronic daily (>10 mg) or alternate daily (>20 mg on alternate days) use of systemic corticosteroids within the 4 weeks prior to Visit 1 (Day -42 to -10) or initiation of any dosage of systemic corticosteroids within 72 hours prior to Visit 2 (Day 1).
3. Use of hydroxychloroquine or immunosuppressants.
4. Initiation of a new antibiotic (oral, intravenous, and/or inhaled) that is not part of the subject's maintenance regimen for treatment of acute respiratory symptoms within 2 weeks prior to screening through Visit 2 (Day 1)
5. Initiation of any new chronic therapy (e.g., Pulmozyme®, hypertonic saline, Kalydeco®, Orkambi®, high-dose ibuprofen azithromycin, TOBI®, Cayston®, nebulized colistiin, bronchodilators, inhaled corticosteroids, etc.) within 4 weeks prior to screening
6. Active treatment for non-tuberculous Mycobacteria
7. History of a sputum culture positive for a Burkholderia cepacia complex organism in the previous 12 months.
8. Current tobacco smoker
9. Oxygen saturation < 92% on room air at Visit 1 (Day -42 to -10)
10. History of pulmonary hypertension
11. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2.5 times the upper limit of normal at screening, documented biliary cirrhosis, or portal hypertension
12. Total bilirubin concentration > 1.2 milligram per deciliter (mg/dL) at screening
13. Creatinine > 1.8 mg/dL at screening
14. Pregnant, breastfeeding, or unwilling to practice birth control between Visit 2 (Day 1) and Telephone Call 3 (Day 56) (acceptable forms of contraception: abstinence, hormonal birth control, intrauterine device, or barrier method plus a spermicidal agent), unless surgically sterilized or postmenopausal
15. Screening hematology with white blood cell count < 4.5 x 109 cells/liter, hematocrit < 30%, and platelets < 150 x 109 platelets/liter
16. History of invasive cancer requiring systemic therapy
17. History of organ transplantation
18. Currently listed for lung transplantation or having potential to be listed for lung transplantation in the succeeding 12 calendar months from screening
19. Subject unlikely to complete the study as determined by the Investigator

Inclusion Criteria for Healthy Volunteer Donors (NOTE: Enrollment for Healthy Volunteers is closed):

1. Male/female age ≥ 18 years to ≤ 40 years
2. Able to understand and sign consent form (a legally authorized representative will not be permitted)

Inclusion Criteria for CF Donors:

1. CF subject enrolled in the main study and consented to this optional procedure

Exclusion Criteria for both Healthy Volunteer (HV) Donors and CF Donors:

1. Fever or current illness on the day of the cell collection
2. Evidence of communicable disease
3. Any significant change in health status within 2 weeks prior to cell collection that the Principal Investigator/Sub-Investigator deems relevant to exclude participation
4. Subject reported history of organ transplantation
5. Subject reported history of human immunodeficiency virus, hepatitis B or C, or syphilis
6. For HV donors only, subject-reported known history of being diagnosed with cystic fibrosis (CF) or being a CF carrier (one copy of CF gene mutation)
7. Positive screening blood test result for any infectious disease.
8. For HV donors only, positive test result for CMV or a CF gene mutation.
9. Pregnant, planning a pregnancy, or breast-feeding at screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2020-08 (Actual); Study Completion 2020-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erica A. Roesch, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ivy SP, Siu LL, Garrett-Mayer E, Rubinstein L. Approaches to phase 1 clinical trial design focused on safety, efficiency, and selected patient populations: a report from the clinical trial design task force of the national cancer institute investigational drug steering committee. Clin Cancer Res. 2010 Mar 15;16(6):1726-36. doi: 10.1158/1078-0432.CCR-09-1961. Epub 2010 Mar 9. PMID 20215542
- [Background] Inamdar AC, Inamdar AA. Mesenchymal stem cell therapy in lung disorders: pathogenesis of lung diseases and mechanism of action of mesenchymal stem cell. Exp Lung Res. 2013 Oct;39(8):315-27. doi: 10.3109/01902148.2013.816803. Epub 2013 Aug 30. PMID 23992090
- [Background] Gebler A, Zabel O, Seliger B. The immunomodulatory capacity of mesenchymal stem cells. Trends Mol Med. 2012 Feb;18(2):128-34. doi: 10.1016/j.molmed.2011.10.004. Epub 2011 Nov 25. PMID 22118960
- [Background] Lalu MM, McIntyre L, Pugliese C, Fergusson D, Winston BW, Marshall JC, Granton J, Stewart DJ; Canadian Critical Care Trials Group. Safety of cell therapy with mesenchymal stromal cells (SafeCell): a systematic review and meta-analysis of clinical trials. PLoS One. 2012;7(10):e47559. doi: 10.1371/journal.pone.0047559. Epub 2012 Oct 25. PMID 23133515
- [Background] Caplan AI. Why are MSCs therapeutic? New data: new insight. J Pathol. 2009 Jan;217(2):318-24. doi: 10.1002/path.2469. PMID 19023885
- [Background] Bonfield TL, Caplan AI. Adult mesenchymal stem cells: an innovative therapeutic for lung diseases. Discov Med. 2010 Apr;9(47):337-45. PMID 20423678
- [Background] Dimarino AM, Caplan AI, Bonfield TL. Mesenchymal stem cells in tissue repair. Front Immunol. 2013 Sep 4;4:201. doi: 10.3389/fimmu.2013.00201. PMID 24027567
- [Background] Antunes MA, Laffey JG, Pelosi P, Rocco PR. Mesenchymal stem cell trials for pulmonary diseases. J Cell Biochem. 2014 Jun;115(6):1023-32. doi: 10.1002/jcb.24783. PMID 24515922
- [Result] Gupta N, Su X, Popov B, Lee JW, Serikov V, Matthay MA. Intrapulmonary delivery of bone marrow-derived mesenchymal stem cells improves survival and attenuates endotoxin-induced acute lung injury in mice. J Immunol. 2007 Aug 1;179(3):1855-63. doi: 10.4049/jimmunol.179.3.1855. PMID 17641052
- [Result] Sutton MT, Fletcher D, Ghosh SK, Weinberg A, van Heeckeren R, Kaur S, Sadeghi Z, Hijaz A, Reese J, Lazarus HM, Lennon DP, Caplan AI, Bonfield TL. Antimicrobial Properties of Mesenchymal Stem Cells: Therapeutic Potential for Cystic Fibrosis Infection, and Treatment. Stem Cells Int. 2016;2016:5303048. doi: 10.1155/2016/5303048. Epub 2016 Jan 26. PMID 26925108

RESULTS

PARTICIPANT FLOW:
Groups:
- 1 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram; 3 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram; 5 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram: One time intravenous infusion of up to 5 x 10^6 allogeneic human mesenchymal stem cells per kilogram body weight (hMSCs/kg). A dose escalation using the "3+3" design was employed. The three doses were 1 x 10^6, 3 x 10^6, and 5 x 10^6 hMSCs/kg. There was no placebo group. All study participants received stem cells.
  Mesenchymal Stem Cells: A single dose, one time infusion (in the vein) of one of the following doses of hMSCs: 1 x 10^6, 3 x 10^6 or 5 x 10^6 hMSCs/kg body weight during Visit 2. A traditional 3+3 design was utilized.
  Allogeneic MSCs were derived from bone marrow aspirates from a healthy donor whose serum tested negative for cytomegalovirus (CMV) antibodies. The healthy donor underwent tests for infectious disease and screening for 41 common cystic fibrosis transmembrane conductance regulator (CFTR) mutations. In addition, the mesenchymal stem cells (MSCs) were validated for in vitro and in vivo efficacy and potency using the in vivo murine pre-clinical model of cystic fibrosis (CF) lung infection and inflammation.
Period: Overall Study
Arm/Group | 1 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram | 3 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram | 5 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram
Started | 3 | 3 | 8
Completed | 3 | 3 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 1 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram; 3 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram; 5 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram: One time intravenous Infusion of up to 5 x 10^6 allogeneic human mesenchymal stem cells per kilogram body weight (hMSCs/kg). A dose escalation using the "3+3" design was employed. The three doses were 1 x 10^6, 3 x 10^6, and 5 x 10^6 hMSCs/kg. There was no placebo group. All study participants received stem cells.
  Mesenchymal Stem Cells (MSCs): A single dose, one time infusion (in the vein) of one of the following doses of hMSCs: 1 x 10^6, 3 x 10^6 or 5 x 10^6 hMSCs/kg body weight during Visit 2. A traditional 3+3 design was utilized.
  Allogeneic MSCs were derived from bone marrow aspirates from a healthy donor whose serum tested negative for cytomegalovirus (CMV) antibodies. The healthy donor underwent tests for infectious disease and screening for 41 common cystic fibrosis transmembrane conductance regulator (CFTR) mutations. In addition, the MSCs were validated for in vitro and in vivo efficacy and potency using the in vivo murine pre-clinical model of cystic fibrosis (CF) lung infection and inflammation.
- Total: Total of all reporting groups
Arm/Group | 1 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram | 3 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram | 5 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram | Total
Number analyzed (Participants) | 3 | 3 | 8 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 8 | 14
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.3 (10.7) | 28.0 (4.7) | 31.7 (12.7) | 30.2 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2 | 4
  Male | 2 | 2 | 6 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 3 | 2 | 8 | 13
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 3 | 8 | 14
Genotype [Count of Participants; unit: Participants] — Number of individuals with two copies of the F508del mutation (F508del homozygous), one copy of the F508del mutation with a different cystic fibrosis causing mutation on the other allele (F508del heterozygous), or two cystic fibrosis causing mutations other than the F508del mutation (other).
  Participants
    F508del Homozygous | 1 | 0 | 3 | 4
    F508del Heterozygous | 1 | 2 | 4 | 7
    Other | 1 | 1 | 1 | 3
Forced Expiratory Volume in the first second (FEV1) % Predicted Distribution [Count of Participants; unit: Participants] — Number of individuals with a Forced Expiratory Volume in the first second (FEV1) percent predicted of less than 70% predicted, between 70-84% predicted, or greater than or equal to 85% predicted. Percent predicted determined using the global lung initiative (GLI). Decreases in FEV1 are associated with more advanced cystic fibrosis lung disease.
  Participants
    <70% | 0 | 2 | 3 | 5
    >=70-84% | 1 | 0 | 2 | 3
    >=85% | 2 | 1 | 3 | 6
Sweat Chloride at Diagnosis [Mean (Standard Deviation); unit: mmol/L] | 107.0 (7.5) | 82.7 (26.6) | 99.4 (20.8) | 97.3 (20.6)
Height [Mean (Standard Deviation); unit: cm] | 167.8 (1.6) | 169.6 (18.7) | 173.6 (8.6) | 171.5 (10.0)
Weight [Mean (Standard Deviation); unit: kg] | 60.1 (13.8) | 63.2 (7.4) | 73.0 (14.1) | 68.2 (13.4)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 21.3 (4.7) | 22.2 (3.3) | 24.3 (4.9) | 23.2 (4.4)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Dose Limiting Toxicity (DLT), Triggered by Occurrence in the First 24 Hours After Human Mesenchymal Stem Cell (hMSC) Infusion of Grade ≥3 Infusion-related Allergic Toxicities
Description: For this study, dose limiting toxicities included the emergence of infusion-related allergic adverse events as well as regimen related toxicities in the first 24 hours after hMSC infusion of a grade ≥ 3 as scored according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. This is the number of participants who experienced a dose limiting toxicity during the study.
Time Frame: 24 hours post infusion
Population: Number of participants with a dose limiting toxicity. All subjects receiving the human mesenchymal stem cell infusing were included.
Measure: Count of Participants; unit: Participants
Groups:
- 1 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram; 3 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram; 5 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram: One time intravenouos Infusion of up to 5 x 10^6 allogeneic human mesenchymal stem cells per kilogram body weight (hMSCs/kg). A dose escalation using the "3+3" design was employed. The three doses were 1 x 10^6, 3 x 10^6, and 5 x 10^6 hMSCs/kg. There was no placebo group. All study participants received stem cells.
  Mesenchymal Stem Cells (MSCs): A single dose, one time infusion (in the vein) of one of the following doses of hMSCs: 1 x 10^6, 3 x 10^6 or 5 x 10^6 hMSCs/kg body weight during Visit 2. A traditional 3+3 design was utilized.
  Allogeneic MSCs were derived from bone marrow aspirates from a healthy donor whose serum tested negative for cytomegalovirus (CMV) antibodies. The healthy donor underwent tests for infectious disease and screening for 41 common cystic fibrosis transmembrane conductance regulator (CFTR) mutations. In addition, the MSCs were validated for in vitro and in vivo efficacy and potency using the in vivo murine pre-clinical model of cystic fibrosis lung infection and inflammation.
Arm/Group | 1 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram | 3 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram | 5 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram
Number analyzed (Participants) | 3 | 3 | 8
Participants | 0 | 0 | 0

2. Primary Outcome: Number of Serious Adverse Events and Number of Non-Serious Adverse Events
Description: Participants were followed for 12 months after human mesenchymal stem cell infusion. All events from the infusion date through the end of follow-up were included. This shows the total number of adverse events or serious adverse events occurring in each dosing cohort.
Time Frame: 1 year
Population: All subjects who received human mesenchymal stem cells were included in the analysis.
Measure: Number; unit: number of adverse events
Arm/Group | 1 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram | 3 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram | 5 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram
Number analyzed (Participants) | 3 | 3 | 8
number of adverse events
  Serious Adverse Event | 3 | 3 | 3
  Non-Serious Adverse Event | 16 | 31 | 68

3. Primary Outcome: Number of Pulmonary Exacerbations Requiring Intravenous Antibiotics
Description: Participants were followed for 12 months after human mesenchymal stem cell infusion. All events occurring from the infusion date through the end of follow-up were included. This shows the number of pulmonary exacerbations requiring intravenous antibiotics in each dosing cohort.
Time Frame: 1 year
Population: All subjects who received human mesenchymal stem cells were included in the analysis.
Measure: Number; unit: pulmonary exacerbations
Arm/Group | 1 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram | 3 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram | 5 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram
Number analyzed (Participants) | 3 | 3 | 8
pulmonary exacerbations | 2 | 3 | 2

4. Primary Outcome: Forced Expiratory Volume in the First Second (FEV1) % Predicted at Baseline and 30 Minutes, 4 Hours, 24 Hours, 7 Days, 14 Days, 28 Days, 3 Months, 6 Months Post Human Mesenchymal Stem Cell Infusion.
Description: Lung function was followed for 6 months post human mesenchymal stem cell infusion. This shows the mean forced expiratory volume in the first second (FEV1) percent predicted for each cohort throughout the study.
Time Frame: Baseline and 30 minutes, 4 hours, 24 hours, 7 days, 14 days, 28 days, 3 months, 6 months Post Human Mesenchymal Stem Cell Infusion
Population: All subjects who received human mesenchymal stem cells were included in the analysis.
Measure: Mean (Standard Deviation); unit: FEV1 percent predicted
Groups:
- 1 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilgoram; 3 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram; 5 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram: One time intravenouos infusion of up to 5 x 10^6 allogeneic human mesenchymal stem cells per kilogram body weight (hMSCs/kg). A dose escalation using the "3+3" design was employed. The three doses were 1 x 10^6, 3 x 10^6, and 5 x 10^6 hMSCs/kg. There was no placebo group. All study participants received stem cells.
  Mesenchymal Stem Cells (MSCs): A single dose, one time infusion (in the vein) of one of the following doses of hMSCs: 1 x 10^6, 3 x 10^6 or 5 x 10^6 hMSCs/kg body weight during Visit 2. A traditional 3+3 design was utilized.
  Allogeneic MSCs were derived from bone marrow aspirates from a healthy donor whose serum tested negative for cytomegalovirus (CMV) antibodies. The healthy donor underwent tests for infectious disease and screening for 41 common cystic fibrosis transmembrane conductance regulator (CFTR) mutations. In addition, the MSCs were validated for in vitro and in vivo efficacy and potency using the in vivo murine pre-clinical model of cystic fibrosis lung infection and inflammation.
Arm/Group | 1 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilgoram | 3 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram | 5 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram
Number analyzed (Participants) | 3 | 3 | 8
FEV1 percent predicted
  FEV1 at baseline | 83.2 (8.5) | 71.4 (13.5) | 77.7 (20.2)
  FEV1 30 minutes post infusion | 79.7 (9.9) | 69.0 (9.6) | 75.3 (20.3)
  FEV1 4 hours post infusion | 83.1 (14.3) | 69.0 (14.2) | 75.2 (21.1)
  FEV1 24 hours post infusion | 86.4 (15.6) | 75.1 (13.7) | 77.4 (21.2)
  FEV1 7 days post infusion | 83.6 (4.3) | 64.5 (9.8) | 76.5 (18.7)
  FEV1 14 days post infusion | 85.6 (8.0) | 67.5 (8.4) | 75.6 (19.9)
  FEV1 28 days post infusion | 85.4 (11.4) | 69.8 (12.0) | 77.8 (19.7)
  FEV1 3 months post infusion | 89.4 (17.2) | 70.9 (14.2) | 76.1 (19.5)
  FEV1 6 months post infusion | 91.3 (18.7) | 70.0 (11.1) | 76.1 (20.7)

5. Secondary Outcome: Serum Inflammatory Markers - Calportectin Measurements at Baseline, Day 7, and Day 28
Description: Serum inflammatory markers including Calprotectin were collected at baseline and at the visits 7 days and 28 days post human mesenchymal stem cell (hMSC) infusion. Mean values with standard deviation are shown. The lower limit for detection for calportectin was 88.3 picogram per millilitre.
Time Frame: Baseline, Day 7, Day 28 post human mesenchymal stem cell infusion
Population: All subjects who received human mesenchymal stem cells were included in the analysis.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | 1 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram | 3 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram | 5 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram
Number analyzed (Participants) | 3 | 3 | 8
pg/ml
  Baseline | 9735.2 (16708.9) | 88.3 (0) | 93.1 (5.1)
  Day 7 | 88.3 (0) | 94.2 (10.2) | 93.1 (5.1)
  Day 28 | 88.3 (0) | 88.3 (0) | 91.1 (5.1)

6. Secondary Outcome: Serum Inflammatory Markers - Granulocyte-Macrophage Colony-Stimulating Factor (GM-CSF) Measurements at Baseline, Day 7, and Day 28
Description: Serum inflammatory markers including Granulocyte-Macrophage Colony-Stimulating Factor (GM-CSF) were collected at baseline and at the visits 7 days and 28 days post human mesenchymal stem cell (hMSC) infusion. Mean values with standard deviation are shown. The lower limit for detection for GM-CSF was 2.6 picograms per milliliter.
Time Frame: Baseline, Day 7, Day 28 post human mesenchymal stem cell infusion
Population: All subjects who received human mesenchymal stem cells were included in the analysis.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | 1 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram | 3 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram | 5 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram
Number analyzed (Participants) | 3 | 3 | 8
pg/ml
  Baseline | 3.3 (1.3) | 3.5 (1.2) | 7.1 (3.1)
  Day 7 | 5.2 (1.5) | 4.3 (0.1) | 6.2 (3.7)
  Day 28 | 4.6 (2.4) | 2.6 (0) | 6.7 (3.3)

7. Secondary Outcome: Serum Inflammatory Markers - Interleukin-1 (IL-1) Measurements at Baseline, Day 7, and Day 28
Description: Serum inflammatory markers including interleukin -1 (IL-1) were collected at baseline and at the visits 7 days and 28 days post human mesenchymal stem cell (hMSC) infusion. Mean values with standard deviation are shown. The lower limit for detection for IL-1 was 13.1 picograms per milliliter.
Time Frame: Baseline, Day 7, Day 28 post human mesenchymal stem cell infusion
Population: All subjects who received human mesenchymal stem cells were included in the analysis.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | 1 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram | 3 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram | 5 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram
Number analyzed (Participants) | 3 | 3 | 8
pg/ml
  Baseline | 15.9 (4.8) | 13.1 (0) | 13.1 (0)
  Day 7 | 13.1 (0) | 13.1 (0) | 13.1 (0)
  Day 28 | 13.1 (0) | 13.1 (0) | 13.1 (0)

8. Secondary Outcome: Serum Inflammatory Markers - Interleukin-17 (IL-17) Measurements at Baseline, Day 7, and Day 28
Description: Serum inflammatory markers including interleukin -17 (IL-17) were collected at baseline and at the visits 7 days and 28 days post human mesenchymal stem cell (hMSC) infusion. Mean values with standard deviation are shown. The lower limit for detection for IL-17 was 13.5 picograms per milliliter.
Time Frame: Baseline, Day 7, Day 28 post human mesenchymal stem cell infusion
Population: All subjects who received human mesenchymal stem cells were included in the analysis.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | 1 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram | 3 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram | 5 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram
Number analyzed (Participants) | 3 | 3 | 8
pg/ml
  Baseline | 13.5 (0) | 13.8 (0.6) | 18.0 (26.7)
  Day 7 | 20.7 (12.6) | 15.7 (3.8) | 18.0 (26.7)
  Day 28 | 22.0 (11.5) | 14.9 (2.5) | 17.3 (24.5)

9. Secondary Outcome: Serum Inflammatory Markers - Interleukin-6 (IL-6) Measurements at Baseline, Day 7, and Day 28
Description: Serum inflammatory markers including interleukin -6 (IL-6) were collected at baseline and at the visits 7 days and 28 days post human mesenchymal stem cell (hMSC) infusion. Mean values with standard deviation are shown. The lower limit for detection for IL-6 was 13.5 picograms per milliliter.
Time Frame: Baseline, Day 7, Day 28 post human mesenchymal stem cell infusion
Population: All subjects who received human mesenchymal stem cells were included in the analysis.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | 1 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram | 3 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram | 5 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram
Number analyzed (Participants) | 3 | 3 | 8
pg/ml
  Baseline | 4.1 (1.6) | 4.6 (2.7) | 4.8 (5.4)
  Day 7 | 2.6 (0.3) | 5.7 (5.9) | 4.6 (4.7)
  Day 28 | 3.1 (0.8) | 3.7 (2.0) | 5.4 (5.5)

10. Secondary Outcome: Serum Inflammatory Markers - Interleukin-8 (IL-8) Measurements at Baseline, Day 7, and Day 28
Description: Serum inflammatory markers including interleukin -8 (IL-8) were collected at baseline and at the visits 7 days and 28 days post human mesenchymal stem cell (hMSC) infusion. Mean values with standard deviation are shown. The lower limit for detection for IL-8 was 13.9 picograms per milliliter.
Time Frame: Baseline, Day 7, Day 28 post human mesenchymal stem cell infusion
Population: All subjects who received human mesenchymal stem cells were included in the analysis.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | 1 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram | 3 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram | 5 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram
Number analyzed (Participants) | 3 | 3 | 8
pg/ml
  Baseline | 2225.6 (3824.4) | 22.9 (15.5) | 24.9 (26.7)
  Day 7 | 21.5 (6.0) | 17.0 (5.4) | 32.7 (35.5)
  Day 28 | 22.9 (7.9) | 18.7 (8.3) | 21.8 (13.6)

11. Secondary Outcome: Serum Inflammatory Markers - Myeloperoxidase (MPO) Measurements at Baseline, Day 7, and Day 28
Description: Serum inflammatory markers including myeloperoxidase (MPO) were collected at baseline and at the visits 7 days and 28 days post human mesenchymal stem cell (hMSC) infusion. Mean values with standard deviation are shown.
Time Frame: Baseline, Day 7, Day 28 post human mesenchymal stem cell infusion
Population: All subjects who received human mesenchymal stem cells were included in the analysis.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | 1 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram | 3 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram | 5 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram
Number analyzed (Participants) | 3 | 3 | 8
pg/ml
  Baseline | 74168.3 (40518.7) | 245158.5 (88431.6) | 245928.3 (122070.0)
  Day 7 | 122043.5 (58466.6) | 305665.3 (85217.9) | 225988.7 (128113.3)
  Day 28 | 93838.6 (26655.9) | 250501.1 (205136.2) | 226155.5 (142171.8)

12. Secondary Outcome: Serum Inflammatory Markers - Tumor Necrosis Factor Alpha (TNF-a) Measurements at Baseline, Day 7, and Day 28
Description: Serum inflammatory markers including tumor necrosis factor alpha (TNF-a) were collected at baseline and at the visits 7 days and 28 days post human mesenchymal stem cell (hMSC) infusion. Mean values with standard deviation are shown. The lower limit of detection for TNF-a was 12.9 picograms per millilter.
Time Frame: Baseline, Day 7, Day 28 post human mesenchymal stem cell infusion
Population: All subjects who received human mesenchymal stem cells were included in the analysis.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | 1 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram | 3 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram | 5 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram
Number analyzed (Participants) | 3 | 3 | 8
pg/ml
  Baseline | 12.9 (0) | 12.9 (0) | 19.5 (6.6)
  Day 7 | 12.9 (0) | 14.2 (2.3) | 19.2 (6.8)
  Day 28 | 12.9 (0) | 12.9 (0) | 19.2 (6.8)

13. Secondary Outcome: Sputum Inflammatory Markers - Granulocyte-Macrophage Colony-Stimulating Factor (GM-CSF) Measurements at Baseline, Day 7, and Day 28
Description: Sputum inflammatory markers including granulocyte-macrophage colony-stimulating factor (GM-CSF) were collected at baseline and at the visits 7 days and 28 days post human mesenchymal stem cell (hMSC) infusion. Mean values with range are shown.
Time Frame: Baseline, Day 7, Day 28 post human mesenchymal stem cell infusion
Population: Only 4 subjects were able to produce sputum at all time points.
Measure: Mean (Full Range); unit: pg/ml
Arm/Group | 1 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram | 3 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram | 5 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram
Number analyzed (Participants) | 0 | 2 | 2
pg/ml
  Baseline |  | 1.796 [1.753 to 1.839] | 1.653 [1.209 to 2.097]
  Day 7 |  | 2.755 [1.624 to 3.885] | 1.481 [1.209 to 1.753]
  Day 28 |  | 2.971 [2.488 to 3.453] | 38.799 [1.209 to 76.388]

14. Secondary Outcome: Sputum Inflammatory Markers - Interleukin-1 (IL-1) Measurements at Baseline, Day 7, and Day 28
Description: Sputum inflammatory markers including interleukin-1 (IL-1) were collected at baseline and at the visits 7 days and 28 days post human mesenchymal stem cell (hMSC) infusion. Mean values with range are shown.
Time Frame: Baseline, Day 7, Day 28 post human mesenchymal stem cell infusion
Population: Only 4 subjects were able to produce sputum at all time points.
Measure: Mean (Full Range); unit: pg/ml
Arm/Group | 1 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram | 3 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram | 5 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram
Number analyzed (Participants) | 0 | 2 | 2
pg/ml
  Baseline |  | 1267.24 [1053.10 to 1481.37] | 907.90 [529.62 to 1286.18]
  Day 7 |  | 916.96 [439.02 to 1394.90] | 2432.30 [753.93 to 4110.67]
  Day 28 |  | 1137.81 [1109.64 to 1165.98] | 2501.65 [2153.39 to 2849.91]

15. Secondary Outcome: Sputum Inflammatory Markers - Interleukin-10 (IL-10) Measurements at Baseline, Day 7, and Day 28
Description: Sputum inflammatory markers including interleukin-10 (IL-10) were collected at baseline and at the visits 7 days and 28 days post human mesenchymal stem cell (hMSC) infusion. Mean values with range are shown.
Time Frame: Baseline, Day 7, Day 28 post human mesenchymal stem cell infusion
Population: Only 4 subjects were able to produce sputum at all time points.
Measure: Mean (Full Range); unit: pg/ml
Arm/Group | 1 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram | 3 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram | 5 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram
Number analyzed (Participants) | 0 | 2 | 2
pg/ml
  Baseline |  | 1.614 [1.614 to 1.614] | 0.979 [0.724 to 1.233]
  Day 7 |  | 1.614 [1.614 to 1.614] | 1.424 [1.233 to 1.614]
  Day 28 |  | 1.614 [1.614 to 1.614] | 1.233 [1.233 to 1.233]

16. Secondary Outcome: Sputum Inflammatory Markers - Interleukin-17 (IL-17) Measurements at Baseline, Day 7, and Day 28
Description: Sputum inflammatory markers including interleukin-17 (IL-17) were collected at baseline and at the visits 7 days and 28 days post human mesenchymal stem cell (hMSC) infusion. Mean values with range are shown.
Time Frame: Baseline, Day 7, Day 28 post human mesenchymal stem cell infusion
Population: Only 4 subjects were able to produce sputum at all time points.
Measure: Mean (Full Range); unit: pg/ml
Arm/Group | 1 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram | 3 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram | 5 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram
Number analyzed (Participants) | 0 | 2 | 2
pg/ml
  Baseline |  | 1.076 [1.019 to 1.132] | 0.752 [0.643 to 0.861]
  Day 7 |  | 1.144 [0.961 to 1.427] | 0.480 [0.318 to 0.643]
  Day 28 |  | 1.167 [0.906 to 1.427] | 0.643 [0.643 to 0.643]

17. Secondary Outcome: Sputum Inflammatory Markers - Interleukin-6 (IL-6) Measurements at Baseline, Day 7, and Day 28
Description: Sputum inflammatory markers including interleukin-6 (IL-6) were collected at baseline and at the visits 7 days and 28 days post human mesenchymal stem cell (hMSC) infusion. Mean values with range are shown.
Time Frame: Baseline, Day 7, Day 28 post human mesenchymal stem cell infusion
Population: Only 4 subjects were able to produce sputum at all time points.
Measure: Mean (Full Range); unit: pg/ml
Arm/Group | 1 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram | 3 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram | 5 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram
Number analyzed (Participants) | 0 | 2 | 2
pg/ml
  Baseline |  | 4.908 [4.837 to 4.979] | 4.253 [4.072 to 4.434]
  Day 7 |  | 4.188 [3.448 to 4.927] | 4.501 [1.640 to 7.362]
  Day 28 |  | 6.733 [4.396 to 9.069] | 4.118 [1.640 to 6.596]

18. Secondary Outcome: Sputum Inflammatory Markers - Interleukin-8 (IL-8) Measurements at Baseline, Day 7, and Day 28
Description: Sputum inflammatory markers including interleukin-8 (IL-8) were collected at baseline and at the visits 7 days and 28 days post human mesenchymal stem cell (hMSC) infusion. Mean values with range are shown.
Time Frame: Baseline, Day 7, Day 28 post human mesenchymal stem cell infusion
Population: Only 4 subjects were able to produce sputum at all time points.
Measure: Mean (Full Range); unit: pg/ml
Arm/Group | 1 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram | 3 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram | 5 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram
Number analyzed (Participants) | 0 | 2 | 2
pg/ml
  Baseline |  | 1814.44 [1508.23 to 2120.64] | 7862.76 [3412.01 to 12313.50]
  Day 7 |  | 2398.03 [2292.14 to 2503.91] | 5061.17 [2592.75 to 7529.59]
  Day 28 |  | 1538.79 [1397.77 to 1679.82] | 9348.03 [8361.68 to 10334.38]

19. Secondary Outcome: Sputum Inflammatory Markers - Macrophage Inflammatory Protein-3 Alpha (MIP-3a) Measurements at Baseline, Day 7, and Day 28
Description: Sputum inflammatory markers including macrophage inflammatory protein-3 alpha (MIP-3a) were collected at baseline and at the visits 7 days and 28 days post human mesenchymal stem cell (hMSC) infusion. Mean values with range are shown.
Time Frame: Baseline, Day 7, Day 28 post human mesenchymal stem cell infusion
Population: Only 4 subjects were able to produce sputum at all time points.
Measure: Mean (Full Range); unit: pg/ml
Arm/Group | 1 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram | 3 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram | 5 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram
Number analyzed (Participants) | 0 | 2 | 2
pg/ml
  Baseline |  | 18.01 [7.78 to 28.23] | 7.78 [7.78 to 7.78]
  Day 7 |  | 16.06 [7.78 to 24.34] | 14.426 [7.78 to 21.07]
  Day 28 |  | 17.03 [7.78 to 26.28] | 7.83 [7.78 to 7.87]

20. Secondary Outcome: Sputum Inflammatory Markers - Tumor Necrosis Factor Alpha (TNF-a) Measurements at Baseline, Day 7, and Day 28
Description: Sputum inflammatory markers including tumor necrosis factor alpha (TNF-a) were collected at baseline and at the visits 7 days and 28 days post human mesenchymal stem cell (hMSC) infusion. Mean values with range are shown.
Time Frame: Baseline, Day 7, Day 28 post human mesenchymal stem cell infusion
Population: Only 4 subjects were able to produce sputum at all time points.
Measure: Mean (Full Range); unit: pg/ml
Arm/Group | 1 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram | 3 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram | 5 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram
Number analyzed (Participants) | 0 | 2 | 2
pg/ml
  Baseline |  | 216.572 [12.591 to 420.553] | 14.606 [13.693 to 15.518]
  Day 7 |  | 45.069 [15.892 to 74.245] | 25.567 [10.2 to 40.933]
  Day 28 |  | 26.858 [11.052 to 42.664] | 21.861 [7.225 to 36.497]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | 1 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram | 3 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram | 5 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/8
Serious Adverse Events (participants affected / at risk) | 2/3 | 2/3 | 2/8
Other Adverse Events (participants affected / at risk) | 2/3 | 2/3 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram (N=3) | 3 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram (N=3) | 5 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram (N=8)
Cystic Fibrosis Pulmonary Exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (3) | 2 (2) — Pulmonary exacerbation requiring hospital admission for IV antibiotics.
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — Constipation requiring admission to the hopsital.
Right Common Iliac Thrombus (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) — Right common iliac thrombus requiring hospital admission.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram (N=3) | 3 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram (N=3) | 5 x 10^6 Human Allogeneic Mesenchymal Stem Cells Per Kilogram (N=8)
Right leg pain (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (2) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (1)
Constipation (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Change in Appetite (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bleeding Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Slow Weight Gain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 2 (2)
Non-cardiac Chest Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Risk of Pathogen Exposure (General disorders) | 1 (1) | 0 (0) | 0 (0)
Febrile Viral Illness (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Upper Respiratory Infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Weight Loss (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Bilateral Lower Extremity Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Body Aches (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Generalized Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Right Heel Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Headahche (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Memory Impairment (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Suicidal Ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Cystoscopy (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Increased Creatinine (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Ureter Stricture (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary Hesitancy (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urology Procedure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Breast Swelling (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Increased Sputum Production (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 3 (3)
Cystic Fibrosis Pulmonary Exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (5) | 3 (4)
Decreased FEV1 (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (3)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (5)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (4)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (2)
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (4)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cold Sore (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Left Buttock Condyloma (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Left Shoulder Cyst Removal (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Mild Pruritus Ani (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Mild Non-Tender, Non-Fluctuant Erythema Around IV Insertion Site (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (2)
Right leg edema (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
PICC Line Insertion (Surgical and medical procedures) | 1 (1) | 0 (0) | 1 (1)
CT Scan of Right Lower Extermity (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Left Popliteal Venogram and Lysis Catheter Placement (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Lysis Catheter Removal (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
PICC Line (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
PICC Line Right Upper Extremity (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Limitations include the small sample size and short study period. The primary objective was to determine safety, therefore therapeutic exposure was limited to a single dose of human mesenchymal stem cells (hMSCs). The clinical trial was not powered to detect changes in secondary exploratory measures, thus limiting our understanding of the impact of hMSCs on inflammation in cystic fibrosis. The ability to assess efficacy was further limited by the inability of participants to produce sputum.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-12-17): https://cdn.clinicaltrials.gov/large-docs/21/NCT02866721/Prot_SAP_000.pdf
  • Informed Consent Form (2020-12-03): https://cdn.clinicaltrials.gov/large-docs/21/NCT02866721/ICF_001.pdf